CLINICAL TRIAL: NCT06516939
Title: The Application of Bovine Basic Fibroblast Growth Factor Gel in the Treatment of Sensitive Skin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Dermatology Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-06
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Sensitive Skin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Application of Bovine Basic Fibroblast Growth Factor Gel (Experimental)
  Interventions: Drug: bFGF
- Bovine Basic Gel (Placebo Comparator)
  Interventions: Drug: Bovine Basic Gel

INTERVENTIONS:
Drug: bFGF — Half-face randomized control
  Arms: The Application of Bovine Basic Fibroblast Growth Factor Gel
Drug: Bovine Basic Gel — Bovine Basic Gel
  Arms: Bovine Basic Gel

SUMMARY:
The Application of Bovine Basic Fibroblast Growth Factor Gel in the Treatment of Sensitive Skin

ELIGIBILITY:
Inclusion Criteria:

1. Sensitive skin with a diagnosis of persistent erythema and a lactate irritation test score of 2-3
2. No related skin care products including bovine alkaline fibroblast growth factor were used within 1 month before participating in the experiment, and photoelectric treatment measures were not carried out
3. Physical sunscreen should be strict during enrollment

Exclusion Criteria:

1. Children
2. Have serious heart, liver, kidney, and blood system diseases, and severe immunocompromise
3. Patients with mental illness or cancer
4. Those who have received glucocorticoids, calcineurin inhibitors, topical small molecule drugs, antibiotics or tretinoin within 3 months
5. Those who are allergic to basic fibroblast growth factor gel and its components
6. Acute dermatitis of the face and perifolliculitis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Estimated)

PRIMARY OUTCOMES:
erythema index | 0、1、2、4 week
  The change rate in lesion clearance of face at 1 month after treatment will be measured as the primary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Skin Disease Hospital, Shanghai, China